CLINICAL TRIAL: NCT01320007
Title: Lung Impedance Monitoring In Treatment of Chronic Heart Failure
Acronym: LIMIT-CHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BLT006957
Record Dates: First submitted 2011-02-21; First posted 2011-03-22 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1: Optivol Group (Experimental)
  Interventions: Drug: Preset increase in frusemide dose
- Group 2: Optivol alarm muted (Active Comparator)
  Interventions: Other: No intervention

INTERVENTIONS:
Drug: Preset increase in frusemide dose — All patients in Group 1 will have the Optivol function and alerts switched on. Optivol levels will be downloaded monthly via the Medtronic Carelink Network (for those patients who have it) or during pacemaker follow up appointments.
  If the Optivol alarm goes off, all patients will be requested to contact a member of the research team by phone and those with rising Optivol (irrespective of the presence or absence of heart failure symptoms) will be requested to increase the dose of diuretic that they are on by 50% for 1 week then revert to their usual dose after 7 days. A routine renal function check will be performed at the end of the week.
  Arms: Group 1: Optivol Group
Other: No intervention — The Optivol data for these patients will be downloaded periodically (at each scheduled device check) and recorded but will not be available at follow up in the heart failure clinic.. These patients will act as controls for group 1 patients. They will undergo baseline investigations and then will undergo routine heart failure treatment and follow-up in the heart failure clinic. These will include a routine clinical evaluation, body weight and blood analysis as per the heart failure clinic protocol. Medications will be reviewed and changed according to clinical needs.
  Arms: Group 2: Optivol alarm muted

SUMMARY:
Heart failure is a major clinical problem that is increasing in magnitude and the cost of management of heart failure is escalating. A significant part of this cost is related to unplanned acute presentation to emergency departments and hospitalisation with worsening shortness of breath due to increased fluid content in the lungs.

Many heart failure patients are already fitted with defibrillators to protect them from the risk of fast heart rhythms and sudden death and are followed up in both the heart failure clinics and defibrillator clinics. Recently some of the defibrillators fitted have been equipped with an extra function that can detect and warn of changes in the fluid content of the lungs very early even before the patient starts to complain of any shortness of breath and before any signs of fluid overload are seen clinically. However, it is not known how to deal with these warnings if they occur very early and it is not known whether a medical intervention at his stage is beneficial to prevent progression and eventual hospital admission. In the majority of cases, early warnings of this kind are ignored or this function is disabled at implantation of the device.

The current study will involve patients who have already been fitted with a device with the above capability. The investigators will use the new function to guide management of these patients and compare their outcome with similar patients who are fitted with devices without it. The investigators will attempt to manage early warnings by a predetermined increase in medications in a group of patients and compare their clinical course to a similar group in whom no action is taken.

ELIGIBILITY:
Inclusion Criteria:

* Previously fitted with an ICD or a CRT-D device for primary or secondary prevention (for at least 34 days) with a Medtronic Optivol capable Device
* Previous hospital admission for decompensated heart failure
* Left ventricular systolic dysfunction (EF <50%)
* Currently compensated heart failure with a functional class of III or better
* All patients will be on optimal medical treatment including a beta blocker, an ACEI (or ARB) and spironolactone unless contraindicated or not tolerated

Exclusion Criteria:

* Decompensated patients who have NYHA class IV or clinical signs of lung congestion at time of evaluation (these patients may be included later if/when their NYHA class improves)
* Patients with a high Optivol fluid index at time of evaluation (these patients may be included later when the Optivol fluid index comes down)
* Patients with advanced renal failure ± dialysis (Chronic Kidney Disease class 4 or 5 with an estimated GFR of <30 ml/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The number of unplanned hospitalisations or acute unscheduled care in the emergency department or heart failure clinic | 1 year
  The primary study end-point will be a comparison between groups 1 and 2 regarding the ratio of the number of readmissions for heart failure to the total number of patients in each group of the two main groups over the course of the study (i.e. number of readmissions per patient)

SECONDARY OUTCOMES:
NYHA functional Class improvement of at least 1 grade | 1 year
  The proportion of patients achieving at least 1 grade improvement in New York Heart Association functional class in each group
Minnesota Quality of Life Score improvement in each group | 1 Year
  A comparison between the 2 study groups regarding the magnitude of improvement in the Minnesota Living with Heart Failure (questionnaire) score at 1 year compared to baseline
Change in the 6 minute walk test(6MWT)distance in metres | 1 year
  A comparison between the change in the 6MWT distance covered (at 1 year compared to baseline) in each of the 2 study groups
Change in the level of BNP in serum (pg/ml) | 1 year
  A comparison between between the 2 study groups regarding the change in level of BNP at 1 year compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Schilling, Md FRCP, Principal Investigator — Barts and the London NHS Trust, Queen Mary University of London
Locations (1):
- St Bartholomew's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Domenichini G, Rahneva T, Diab IG, Dhillon OS, Campbell NG, Finlay MC, Baker V, Hunter RJ, Earley MJ, Schilling RJ. The lung impedance monitoring in treatment of chronic heart failure (the LIMIT-CHF study). Europace. 2016 Mar;18(3):428-35. doi: 10.1093/europace/euv293. Epub 2015 Dec 18. PMID 26683599